CLINICAL TRIAL: NCT03716479
Title: The Effect of Gum Acacia on Satiety, Glycemic Response and Gastrointestinal Tolerance
Brief Title: Gum Acacia and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00004203
Record Dates: First submitted 2018-08-29; First posted 2018-10-23 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Diet Modification

STUDY DESIGN:
Intervention Model Description: subjects will consume 0, and 2 doses of acacia gum
Who Masked: Participant, Investigator
Masking Description: fiber will be mixed into orange juice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 fiber (Experimental): 0 grams fiber added to orange juice
  Interventions: Other: Placebo/Control
- low fiber (Experimental): 20 grams of acacia gum added to orange juice
  Interventions: Other: Low Fiber
- high fiber (Experimental): 40 grams of acacia gum added to orange juice
  Interventions: Other: High Fiber

INTERVENTIONS:
Other: Low Fiber — 20 g of acacia gum will be added to orange juice
  Arms: low fiber
Other: High Fiber — 40 g of acacia gum will be added to orange juice
  Arms: high fiber
Other: Placebo/Control — No acacia gum will be added to orange juice.
  Arms: 0 fiber

SUMMARY:
This study will provide needed insight on the satiety and blood glucose and l effects of the soluble fiber gum acacia at 20g and 40g doses.

DETAILED DESCRIPTION:
This is a randomized, single-blind, crossover, intervention study testing the satiety and blood glucose effects of the soluble fiber gum acacia.

ELIGIBILITY:
Inclusion Criteria: BMI between 18 and 29 kg/m2

Exclusion Criteria:

* distaste for bagels and cream cheese, orange juice or cheese pizza;
* current smoker;
* restrained eating habits;
* recent weight change;
* any history of disease or significant past medical history;
* are vegetarian;
* do not normally eat breakfast or lunch;
* pregnant or lactating;
* irregular menstrual cycles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | 0, 30, 60, 120, 180, and 240 minutes after breakfast; Area under the curve (AUC) will be calculated for each treatment
  Blood will be taken via finger stick
Appetite Sensation | 15, 30, 45, 60, 90, 120, 180 and 240 minutes after breakfast; Area under the curve (AUC) will be calculated for each treatment
  Subjective visual analog scale (VAS) will be utilized to assess hunger, fullness and desire to eat

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No